CLINICAL TRIAL: NCT06168942
Title: Laminar Left Atrial Appendage Elimination (LAAX) Pivotal IDE Study
Brief Title: A Pivotal Investigational Device Exemption Study on Laminar Left Atrial Appendage Elimination
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Potential unwrapping of the LAA post implant with clinically significant leaks.
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAM202403; LAM202403 (Other: Biosense Webster, Inc.); CL-0059 (Other: Laminar, Inc.)
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Non-valvular Atrial Fibrillation; Stroke; Systemic Embolism
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Laminar Device (Experimental): Participants will be treated with the Laminar Left Atrial Appendage Closure System.
  Interventions: Device: Experimental: Laminar Left Atrial Appendage Closure System
- Control left atrial appendage closure (LAAC) (Active Comparator): Participants will be treated with a commercially-available LAAC device.
  Interventions: Device: Active Comparator: WATCHMAN / Amulet

INTERVENTIONS:
Device: Experimental: Laminar Left Atrial Appendage Closure System — Treatment with the Laminar Left Atrial Appendage Closure System.
  Arms: Laminar Device
Device: Active Comparator: WATCHMAN / Amulet — Treatment with a WATCHMAN left atrial appendage closure device / Amulet left atrial appendage occluder.
  Arms: Control left atrial appendage closure (LAAC)

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of Laminar Left Atrial Appendage Closure (LAAC) device as compared to the commercially available LAAC devices in participants with non-valvular atrial fibrillation (NVAF) to reduce the risk of stroke (blocked blood vessel or bleeding in brain) and systemic embolism (blockage in a blood vessel harming vital organs).

DETAILED DESCRIPTION:
This prospective, randomized, controlled, multicenter, open-label pivotal clinical study will enroll participants with non-valvular atrial fibrillation who are eligible for short-term anticoagulation therapy but have a rationale to seek non-pharmacologic alternative. Participants will be randomized 1:1 to the Laminar Left Atrial Appendage Closure System or commercially available device (WATCHMAN™ left atrial appendage closure device / Amulet™ left atrial appendage occluder).

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of paroxysmal, persistent, or permanent non-valvular atrial fibrillation (NVAF)
* CHA2DS2-VASc score greater than or equal to (>=) 2 in men and >= 3 in women
* Deemed to be clinically indicated for left atrial appendage (LAA) closure by the Site Investigator and a clinician not a part of the procedural team using an evidence-based decision-making tool in accordance with standard of care
* Recommended for chronic oral anticoagulation therapy (OAC) but has an appropriate rationale to seek a non-pharmacologic alternative
* Eligible for the protocol-specified post-procedural antithrombotic regimen
* Willing and able to comply with the protocol, and has provided written informed consent (participant or legally authorized representative) per institutional review board (IRB) requirements

Exclusion Criteria:

* Single episode, transient, or reversible atrial fibrillation (AF) (example, secondary to thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
* Prior cardiac surgery or any procedure that involved pericardial access
* Stage IV kidney disease or Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) less than (<) 30 milliliters per minute per (mL/min)/1.73 square meters (m^2) or participants with end stage renal disease who are dialysis dependent
* Any cardiac or non-cardiac interventional or surgical procedures within 60 days prior to or any planned general surgery, cardiac surgery, or interventional procedure within 60 days after implant (including, but not limited to cardioversion, percutaneous coronary intervention (PCI), cardiac ablation, cataract surgery)
* Left atrial appendage anatomy which cannot accommodate either commercially available control device or the laminar implant per manufacturer instructions for use (IFU) (that is, the anatomy and sizing must be appropriate for a control and the Laminar device to be enrolled in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2032-02-29 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | Up to 12 months
  Composite rate of all-cause mortality will be reported.
Number of Participants With Major Bleeding According to the Bleeding Academic Research Consortium (BARC) Type III or V | Up to 12 months
  The number of participants with major bleeding, according to the BARC type III or V, will be reported.
  Type III
  1. Type IIIa includes overt bleeding plus a hemoglobin drop of 3 to less than (<) 5 grams per deciliter (g/dL) related to bleeding and any transfusion with overt bleeding.
  2. Type IIIb involves overt bleeding plus a hemoglobin drop of greater than or equal to (>=) 5 g/dL related to bleeding, cardiac tamponade, bleeding requiring surgical intervention for control, or bleeding requiring intravenous vasoactive agents.
  3. Type IIIc includes intracranial hemorrhage, with subcategories confirmed by autopsy, imaging, or lumbar puncture, as well as intraocular bleeding compromising vision.
  Type V
  1. Type Va: Probable fatal bleeding; no autopsy or imaging confirmation but clinically suspicious.
  2. Type Vb: Definite fatal bleeding; overt bleeding or autopsy or imaging confirmation.
Number of Participants With Pericardial Effusion Requiring Drainage | Up to 12 months
  Participants with pericardial effusion requiring drainage will be reported. Pericardial effusion is defined as 1) Clinically non-relevant: requiring no intervention, treated pharmacologically and 2) Clinically relevant: treated with therapeutic intervention (pericardiocentesis, surgical intervention, blood transfusion) and/or result in shock or death.
Number of Participants With Device Embolization | Up to 12 months
  Participants with device embolization will be reported. Device embolization is defined as movement of a medical device to an unintended location within the body with resulting obstruction of an organ or vessel.
Number of Participants With Device or Procedure-Related Events Requiring Open Cardiac Surgery or Major Endovascular Intervention | Up to 12 Months
  Participants with device or procedure-related events requiring open cardiac surgery or major endovascular intervention will be reported.
Number of Participants Reporting Ischemic Stroke or Systemic Embolism | Up to 18 Months
  Participant reporting ischemic stroke or systemic embolism will be reported. Systemic embolism is defined as acute vascular insufficiency or occlusion of the extremities or any non-CNS organ associated with clinical, imaging, surgical/autopsy evidence of arterial occlusion in the absence of other likely mechanism (example; trauma, atherosclerosis, or instrumentation).

SECONDARY OUTCOMES:
Number of Participants With Peri-Device Flow | Up to 12 Months
  Peri-Device flow is defined as >= 3 mm in width which communicates beyond the device into the body of the left atrial appendage) per transesophageal echocardiogram (TEE) evaluated by independent core laboratory.
Rate of Device-Related Thrombosis | Up to 12 Months
  Device related thrombosis is defined as density attached to the implanted LAAC device in echocardiographic or computer tomography imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Saibal Kar, MD, Principal Investigator — Los Robles Health System; Devi Nair, MD, Principal Investigator — St. Bernards Heart and Vascular Center
Locations (70):
- United States (44):
  - Grandview Medical Center, Birmingham, Alabama
  - Arizona Arrhythmia Research Group Phoenix Cardio Research Group PCRG, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - OC Medical Center, Fountain Valley, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford Health Care, Palo Alto, California
  - Univeristy of California Davis Health, Rancho Cordova, California
  - Scripps Health, San Diego, California
  - Providence Saint John's Health Center and the Pacific Heart Institute, Santa Monica, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - NCH Healthcare, North Naples, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - The Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Ascension via Christi Hospitals Wichita Inc, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Englewood Health, Englewood, New Jersey
  - Northwell Health, Bay Shore, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University in the City of New York and The New York and Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Bethesda North Hospital Trihealth, Cincinnati, Ohio
  - Lindner Clinical Trial Center/Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Ohio Health, Columbus, Ohio
  - Trident Medical Center, North Charleston, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Texas Heart Institute, Houston, Texas
  - Baylor Scott & White Research Institute at The Heart Hospital Baylor Plano, Plano, Texas
  - Heart Rhythm Associates, Shenandoah, Texas
  - Swedish Medical Center, Seattle, Washington
  - St Joseph Hospital and Medical Center, Tacoma, Washington
  - Mercy Hospital, Janesville, Wisconsin
- Belgium (4):
  - AZORG campus Aalst Moorselbaan, Aalst
  - AZ Sint Jan Brugge Oostende AV, Bruges
  - C.H.U. Brugmann, Brussels
  - CHU Charleroi Chimay, Charleroi
- Nemocnice na Homolce, Prague, Czechia
- Rigshospitalet Copenhagen University Hospital, Copenhagen, Denmark
- France (2):
  - Hopital Prive Jacques Cartier, Massy
  - Clinique Pasteur, Toulouse
- Germany (4):
  - MVZ CCB Frankfurt und Main Taunus GbR, Frankfurt a.M.
  - CVC CardioVascular Center Frankfurt, Frankfurt am Main
  - Asklepios Klinik St. Georg, Hamburg
  - Asklepios Klinik Altona, Hamburg
- Italy (4):
  - Fondazione Toscana Gabriele Monasterio CNR, Massa
  - Centro Cardiologico Monzino, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Policlinico Tor Vergata, Roma
- Vilnius University Hospital Santaros Clinics, Vilnius, Lithuania
- Netherlands (2):
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Erasmus MC, Rotterdam
- Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan, Poland
- Spain (6):
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Clinico San Carlos, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hosp. Alvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No